CLINICAL TRIAL: NCT04766892
Title: An Exploratory, Open-label, Proof-of-concept, Phase 2a Study of Mavacamten (MYK-461) in Participants With Heart Failure With Preserved Ejection Fraction (HFpEF) and Chronic Elevation of Cardiac Biomarkers
Brief Title: A Study of Mavacamten in Participants With HFpEF and Elevation of NT-proBNP With or Without Elevation of cTnT
Acronym: EMBARK-HFpEF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV027-005
Record Dates: First submitted 2021-02-16; First posted 2021-02-23 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: HFpEF; NT-proBNP; Cardiac troponin T
MeSH Terms: conditions — Cardiomyopathy, Familial Restrictive, 3 | interventions — MYK-461

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- mavacamten (MYK-461) (Experimental)
  Interventions: Drug: mavacamten

INTERVENTIONS:
Drug: mavacamten — mavacamten capsules

SUMMARY:
This is a Phase 2a proof-of-concept study to assess safety, tolerability, and preliminary efficacy of mavacamten treatment on biomarker levels in participants with heart failure with preserved ejection fraction (HFpEF) and elevation of NT-proBNP with or without elevation of cTnT. Data from this study will inform future study designs of mavacamten in patients with HFpEF.

ELIGIBILITY:
Key Inclusion Criteria:

1. Is at least 50 years old at Screening.
2. Body weight is greater than 45 kg at Screening.
3. Documented prior objective evidence of heart failure as shown by 1 or more of the following criteria:

   * Previous hospitalization for heart failure with documented radiographic evidence of pulmonary congestion.
   * Elevated LV end-diastolic pressure or pulmonary capillary wedge pressure at rest (≥15 mm Hg) or with exercise (≥25 mm Hg).
   * Elevated level of NT-proBNP (>400 pg/mL) or brain natriuretic peptide (BNP) (>200 pg/mL).
   * Echocardiographic evidence of medial E/e' ratio ≥ 15 or left atrial enlargement (left atrial volume index >34 mL/m2) together with chronic treatment with spironolactone, eplerenone, or a loop diuretic.
4. Meets 1 or more of the following criteria:

   1. A screening hs-cTnT ≥ 99th percentile AND a screening NT-proBNP > 200 pg/mL (if not in atrial fibrillation or atrial flutter) or > 500 pg/mL (if in atrial fibrillation or atrial flutter) OR if the screened participant is of African descent or has a body mass index (BMI) ≥ 30.0 kg/m2, a screening hs-cTnT ≥ 99th percentile, AND a screening NT-proBNP > 160 pg/mL (if not in atrial fibrillation or atrial flutter) or > 400 pg/mL (if in atrial fibrillation or atrial flutter).
   2. A screening NT-proBNP > 300 pg/mL (if not in atrial fibrillation or atrial flutter) or > 750 pg/mL (if in atrial fibrillation or atrial flutter) OR if the screened participant is of African descent or has a BMI ≥ 30.0 kg/m2, a screening NT-proBNP > 240 pg/mL (if not in atrial fibrillation or atrial flutter) or > 600 pg/mL (if in atrial fibrillation or atrial flutter).
5. Has documented LVEF ≥60% at the Screening visit and no history of prior LVEF ≤ 45%.
6. Has maximal left ventricular wall thickness ≥12 mm OR documented elevated left ventricular mass index by 2-dimensional imaging (>95 g/m2 if female and >115 g/m2 if male).
7. Has high quality TTEs without or with echocardiographic contrast agents.
8. Has NYHA class II or III symptoms at Screening.

Key Exclusion Criteria:

1. Has a prior diagnosis of HCM OR a known infiltrative or storage disorder causing HFpEF and/or cardiac hypertrophy, such as amyloidosis, Fabry disease, or Noonan syndrome with LV hypertrophy OR a positive serum immunofixation result.
2. Has a history of syncope within the last 6 months or sustained ventricular tachycardia with exercise within the past 6 months.
3. Has a history of resuscitated sudden cardiac arrest at any time or known appropriate implantable cardioverter defibrillator discharge within 6 months prior to Screening.
4. Has persistent or permanent atrial fibrillation not on anticoagulation for at least 4 weeks prior to Screening and/or is not adequately rate controlled within 6 months prior to Screening.
5. Currently treated or planned treatment during the study with either: (a) a combination of beta blocker and verapamil or a combination of beta blocker and diltiazem, (b) disopyramide, or (c) biotin or biotin-containing supplements/multivitamins.
6. Has known moderate or severe aortic valve stenosis, hemodynamically significant mitral stenosis, or severe mitral or tricuspid regurgitation at Screening.
7. Has severe chronic obstructive pulmonary disease, or other severe pulmonary disease, requiring home oxygen, chronic nebulizer therapy, chronic oral steroid therapy or hospitalized for pulmonary decompensation within 12 months.
8. Has body mass index ≥45.0 kg/m2.
9. Has left ventricular global longitudinal strain by TTE in the range from 0 to -12.0 (assessed by the central laboratory).
10. Has NT-proBNP at Screening >2000 pg/mL.
11. Has acute decompensated heart failure events requiring intravenous (IV) diuretics, IV inotropes, IV vasodilators, or a left ventricular assist device within 30 days prior to Screening.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (21):
- United States (20):
  - Local Institution - 0028, Birmingham, Alabama
  - Local Institution - 0019, Phoenix, Arizona
  - Local Institution - 0011, Tucson, Arizona
  - Local Institution - 0005, Los Angeles, California
  - Local Institution - 0026, San Francisco, California
  - Local Institution - 0020, Jacksonville, Florida
  - Local Institution - 0014, Miami, Florida
  - Local Institution - 0018, Atlanta, Georgia
  - Local Institution - 0004, Chicago, Illinois
  - Local Institution - 0023, Hazel Crest, Illinois
  - Local Institution - 0017, Slidell, Louisiana
  - Local Institution - 0007, Grand Rapids, Michigan
  - Local Institution - 0012, New York, New York
  - Local Institution - 0003, Durham, North Carolina
  - Local Institution - 0016, Oklahoma City, Oklahoma
  - Local Institution - 0010, Portland, Oregon
  - Local Institution - 0001, Portland, Oregon
  - Local Institution - 0002, Philadelphia, Pennsylvania
  - Local Institution - 0008, Charleston, South Carolina
  - Local Institution - 0006, Salt Lake City, Utah
- Local Institution - 0034, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Shah SJ, Rigolli M, Javidialsaadi A, Patel RB, Khadra S, Goyal P, Little S, Wever-Pinzon O, Owens AT, Skali H, Arora P, Solomon SD. Cardiac Myosin Inhibition in Heart Failure With Normal and Supranormal Ejection Fraction: Primary Results of the EMBARK-HFpEF Trial. JAMA Cardiol. 2025 Feb 1;10(2):170-175. doi: 10.1001/jamacardio.2024.3810. PMID 39347697
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 30 participants enrolled and treated
Groups:
- Mavacamten: Mavacamten
Period: Overall Study
Arm/Group | Mavacamten
Started (Started = Treated) | 30
Safety Population | 30
Intent to Treat Population | 30
Completed | 24
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 3
Not completed — Left ventricular ejection fraction (LVEF) Criteria Met | 1

BASELINE CHARACTERISTICS:
Arm/Group | Mavacamten
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.0 (7.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 26
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Treatment-emergent Adverse event (TEAE) is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product; it does not necessarily have to have a causal relationship with this treatment.
Time Frame: From the first dose of study drug through 56 days following last dose of study drug (assessed for an average of 225 days up to a max of approximately 270 days)
Population: Safety Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamten
Number analyzed (Participants) | 30
Participants | 23

2. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: Adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product; it does not necessarily have to have a causal relationship with this treatment. AEs of special interest include: Symptomatic overdose, teratogenicity, and LVEF ≤30%
Time Frame: as for outcome 1
Population: Safety Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamten
Number analyzed (Participants) | 30
Participants
  Symptomatic Overdose | 0
  Outcomes of Pregnancy | 0
  Left Ventricular Ejection Fraction (LVEF) ≤30% | 0

3. Primary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (TESAEs)
Description: Treatment-emergent serious adverse event (TESAE) is defined as any untoward medical occurrence at any dose that: Results in death, Is immediately life-threatening (places the participant at immediate risk of death from the event as it occurred), Requires inpatient hospitalization or prolongation of existing hospitalization, Results in persistent or significant disability or incapacity or substantial disruption of the ability to conduct normal life functions, Results in a congenital abnormality or birth defect, Is an important medical event that may not result in death, be life-threatening, or require hospitalization, but may be considered an SAE when, based upon appropriate medical judgment, it may require medical or surgical intervention to prevent any of the outcomes listed above.
Time Frame: as for outcome 1
Population: Safety Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamten
Number analyzed (Participants) | 30
Participants | 5

4. Primary Outcome: Number of Participants With Laboratory Abnormalities Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: Blood samples were collected to assess the abnormalities in laboratory parameters.
Time Frame: as for outcome 1
Population: Safety Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamten
Number analyzed (Participants) | 30
Participants | 4

5. Primary Outcome: Number of Participants With Abnormal Vital Signs Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Safety Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamten
Number analyzed (Participants) | 30
Participants | 4

6. Primary Outcome: Number of Participants With Cardiac Rhythm Abnormalities Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Safety Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamten
Number analyzed (Participants) | 30
Participants | 5

7. Primary Outcome: Ratio to Baseline at Week 26 in Resting N-Terminal Pro B-Type Natriuretic Peptide (NT-proBNP) Levels
Description: Ratio to baseline in N-terminal pro B-type natriuretic peptide levels.
  The baseline value is defined as the last available value before the first administration of study drug.
Time Frame: At Week 26
Population: All Intention-To-Treat Participants
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Mavacamten
Number analyzed (Participants) | 30
Ratio | 0.7354 [0.5612 to 0.9637]

8. Primary Outcome: Ratio to Baseline at Week 26 in Resting High Sensitivity Cardiac Troponin T (Hs-cTnT) Levels Assessed by High-Sensitivity Assay
Description: Ratio to Baseline in resting high sensitivity cardiac troponin T (hs-cTnT) levels.
  The baseline value is defined as the last available value before the first administration of study drug.
Time Frame: At Week 26
Population: All Intention-To-Treat Participants
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Mavacamten
Number analyzed (Participants) | 30
Ratio | 0.8645 [0.7711 to 0.9693]

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from first dose of study drug until their study completion (assessed up to approximately 1063 days) SAEs and Other AEs were assessed from first dose to 56 days following last dose of study drug (assessed for an average of 225 days up to a max of approximately 270 days)
Description: All-Cause Mortality, Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
  Pre-specified for all doses to be collected combined per treatment.
Arm/Group | Mavacamten
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 5/30
Other Adverse Events (participants affected / at risk) | 18/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mavacamten (N=30)
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Eye haemorrhage (Eye disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal impairment (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mavacamten (N=30)
Atrial flutter (Cardiac disorders) | 2
Asthenia (General disorders) | 2
COVID-19 (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 4
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT04766892/Prot_SAP_000.pdf